CLINICAL TRIAL: NCT00723853
Title: REACH-OUT: Chicago Children's Diabetes Prevention Program
Acronym: REACH-OUT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 11113B
Record Dates: First submitted 2008-07-25; First posted 2008-07-29 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Obesity; Type 2 Diabetes
Keywords: Obesity; Type 2 diabetes; African American children; African American youth; Community based; Family oriented; Obesity & Risk of type 2 diabetes
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2 | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): Reach-Out Program, Nutritional and Exercise Intervention
  Interventions: Behavioral: Reach-Out Program, nutritional and exercise program
- Group 2 (Active Comparator): Reach-In Program, Standard of Care
  Interventions: Behavioral: Reach-Out Program, nutritional and exercise program; Behavioral: Reach-In Program, standard of care

INTERVENTIONS:
Behavioral: Reach-Out Program, nutritional and exercise program — This group will participate in the Reach-Out nutritional and exercise program. This includes 14 weekly, group sessions involving both parents and children.
  During these sessions, participants will receive hands-on education regarding food and exercise habits. Sample nutrition activities include learning to read nutrition labels on foods, a tour of a grocery store and practicing a recipe substituting low fat for high fat ingredients. Exercise activities involve physical activities appropriate for children and adults, respectively. Session leaders will help subjects set personal goals in the areas of nutrition and physical activity, and follow up on subjects' progress each week at sessions and with telephone calls between sessions. At the end of the 14-week program, subjects will be asked to attend four bi-monthly and 18 monthly follow-up sessions in which subjects will continue to meet as a group to work on goals in the areas of nutrition and exercise.
Behavioral: Reach-In Program, standard of care — This group will received standard medical care for their health condition. This includes meeting individually with a dietician to learn about diet, exercise and diabetes. This also includes developing an individualized meal plan.
  Arms: Group 2

SUMMARY:
The purpose of this research study is to evaluate two nutrition and exercise programs in children ages 9-12 who are at risk for developing type 2 diabetes. This study also includes the involvement of parents or guardians who are willing to participate in these programs with the child.

DETAILED DESCRIPTION:
This is a prevention study that evaluates a community-based, family oriented intervention called Reach-Out. The University of Chicago will partner with community organizations including the Women, Infants and Children [WIC] Clinic at the Chicago Department of Public Health Roseland Clinic, South Side YMCA, the Chicago Park District and the Southside Faith-Based Wellness Network of churches to deliver the intervention. Families will be recruited from the high risk population of patients in the University of Chicago Diabetes database and the Chicago Childhood Diabetes Registry; and La Rabida Children's Hospital; and from the broader south side African-American community ("outreach" population). Families will be randomized to behavioral intervention (Reach-Out Program, hands on nutrition and exercise) or control group(Reach-In Program, standard of care consultation).

All who participate in this study will be seen at the University of Chicago GCRC (General Clinical Research Center). They will be asked to come in at the beginning of the study, after 14 weeks, afer 1 year and after 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Overweight (>85th percentile BMI for age and gender) African American child age 9-12 with family history of type 2 diabetes in a first or second degree relative. Parents are secondary subjects.

Exclusion Criteria:

* Inability to give informed consent or unwillingness to be randomized
* Prior diagnosis of diabetes in the child planning to participate
* Pregnancy (women who become pregnant during the study will be omitted from the analysis. Pregnant women will not participate in the exercise sessions).
* Uncontrolled hypertension (SBP> 160 or DBP>100) (JNC V, 1993)
* Uncontrolled dyslipidemia by NCEP III criteria (NCEP, 2001)
* Evidence of significant cardiovascular, pulmonary disease, or other serious illness
* Evidence of alcohol or drug abuse (identified by self-report)
* Musculoskeletal disease serious enough to prevent participation in exercise sessions
* Known or suspected major psychiatric disorder
* Inability to participate in aerobic exercise activities
* Inability to comply with a calorie or fat restricted diet
* Age over 65 years

Ages: 9 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2008-04; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Measure of body habitus (height, weight, waist and hip circumference, body fat by BIE) | 14 weeks, 1 year, 2 years
Biochemical markers (glucose tolerance, lipid panel, insulin, hemoglobin A-1-C) | 14 weeks, 1 year, 2 years

SECONDARY OUTCOMES:
Behavior measurements (food, physical activity, weigh loss, stress, support and television viewing) | 14 weeks, 1 year, 2 years
Cost Assessment (costs incurred to attend meetings, eat healthier, exercise more) | At two weekly meetings

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Burnet, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago GCRC (General Clinical Research Center), Chicago, Illinois, United States